CLINICAL TRIAL: NCT00017433
Title: Phase II Study of Arsenic Trioxide in Patients With Multiple Myeloma
Brief Title: Arsenic Trioxide in Treating Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Purpose: Treatment
Other Study IDs: CTI-1057; CDR0000068688 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-06-06; First posted 2004-01-08 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have relapsed or refractory stage II or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of patients with relapsed or refractory stage II or III multiple myeloma treated with arsenic trioxide. II. Determine the overall and relapse-free survival rates of patients treated with this drug. III. Determine the safety profile of this drug in these patients.

OUTLINE: Patients receive arsenic trioxide IV on days 1-5 and 8-12. Treatment repeats every 4 weeks for up to 6 courses. Patients are followed at 4 weeks after the last treatment dose.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of multiple myeloma Stage II or III (Durie-Salmon) Relapsed or refractory to conventional therapy No monoclonal gammopathy or indolent or smoldering myeloma Measurable disease by serum and urine M protein and/or plasmacytoma

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 70-100% Life expectancy: 3 months Hematopoietic: Granulocyte count greater than 1,200/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 10 g/dL Hepatic: Bilirubin less than 2 times upper limit of normal (ULN) SGOT/SGPT less than 2 times ULN Renal: Creatinine no greater than 2.5 mg/dL Cardiovascular: Absolute QT interval less than 460 msec in the presence of normal potassium and magnesium levels

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 28 days since prior biologic therapy Chemotherapy: No more than 3 prior chemotherapy regimens, including no more than 2 cytotoxic regimens AND 1 high-dose cytotoxic regimen as part of stem cell transplantation Endocrine therapy: At least 28 days since prior endocrine therapy Radiotherapy: At least 28 days since prior radiotherapy (except for focal radiotherapy for symptom control) Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01 (Actual); Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Paradise, MD, Study Chair — CTI BioPharma
Locations (6):
- United States (6):
  - Scripps Clinic, La Jolla, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgia Cancer Specialist, Marietta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Swedish Cancer Institute, Seattle, Washington